CLINICAL TRIAL: NCT06409910
Title: A Phase II Randomized Trial: ALTERNATE DAY ULTRAHYPOFRACTIONATED OR DAILY MODERATELY HYPOFRACTIONATED POST OPERATIVE RADIOTHERAPY
Brief Title: ALTERNATE DAY ULTRAHYPOFRACTIONATED OR DAILY MODERATELY HYPOFRACTIONATED POST OPERATIVE RADIOTHERAPY (AMPORA)
Acronym: AMPORA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-5813
Record Dates: First submitted 2024-03-15; First posted 2024-05-10 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Post-Operative Prostate Cancer
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: Arm 1: External beam radiotherapy 54 Gy in 20 fractions to prostate bed +/- 44 Gy in 20 fractions to pelvic lymph nodes delivered daily.
  Arm 2: External beam radiotherapy 30 Gy in 5 fractions to prostate bed +/- 25 Gy in 5 fractions to pelvic lymph nodes delivered on alternate days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Moderately Hypofractionated Radiotherapy (Experimental): External beam radiotherapy 54 Gy in 20 fractions to prostate bed +/- 44 Gy in 20 fractions to pelvic lymph nodes delivered daily.
  Interventions: Radiation: Radiotherapy
- Arm 2: Ultrahypofractionated Radiotherapy (Experimental): External beam radiotherapy 30 Gy in 5 fractions to prostate bed +/- 25 Gy in 5 fractions to pelvic lymph nodes delivered on alternate days.
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Non-institutional-standard radiotherapy

SUMMARY:
This is a multi-institution, randomized, non-inferiority Phase II trial comparing external beam radiotherapy delivered as 54 Gy in 20 fractions to prostate bed +/- 44 Gy in 20 fractions to pelvic lymph nodes delivered daily with external beam radiotherapy delivered as 30 Gy in 5 fractions to prostate bed +/- 25 Gy in 5 fractions to pelvic lymph nodes delivered on alternate days.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Able to provide informed consent
3. Histologic diagnosis of prostate adenocarcinoma
4. ECOG performance status 0-1
5. Previous radical prostatectomy > 6 months prior to radiotherapy start date
6. Planned to receive post-operative radiation

Exclusion Criteria:

1. Prior pelvic radiotherapy
2. Contraindications to radiotherapy
3. Mets confirmed as per (if scan has been done for clinical care)
4. Participants with visible disease in the prostate bed or pelvic lymph nodes on imaging are not eligible for treatment on study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2030-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Rates of Acute Toxicity | 2 years
  Acute grade ≥2 gastrointestinal toxicity (CTCAE v5.0)

SECONDARY OUTCOMES:
Rates of Acute and Late Toxicity | 2 years
  Acute grade ≥2 genitourinary toxicity (CTCAE v5.0)
Quality of Life Outcomes | 2 years
  EPIC-26 Questionnaire
Quality of Life Outcomes | 2 years
  IPSS Questionnaire
Biochemical disease-free survival | 2 years
  Defined as survival until evidence of either biochemical progression (defined as a rise in prostate-specific antigen (PSA) ≥0.2ng/ml above the PSA nadir followed by a sequentially equal or higher value) following postoperative radiotherapy, clinical or radiological progression, initiation of non-protocol systemic therapy, or death from prostate cancer
Disease Control Rate | 2 years
  Radiographic and/or histopathological disease control rate

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network - Princess Margaret Cancer Centre, Toronto, Ontario, Canada